CLINICAL TRIAL: NCT01838538
Title: Clinical Study in Treatment of Malignant Ascites of Ovarian Cancer With Intraperitoneal Injection Bevacizumab Combined With Intraperitoneal Hyperthermic Perfusion Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, DuNan, Chief Physician, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25396
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Ovarian Cancer With Malignant Ascites
MeSH Terms: interventions — Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab+TC (Experimental): The treatment group were accepted intraperitoneal injection with bevacizumab (avastin) 300mg after each intraperitoneal hyperthermic perfusion chemotherapy for 6 weeks.
  Interventions: Drug: Bevacizumab; Drug: TC:paclitaxel + carboplatin
- TC (Active Comparator): patients were treated with TC chemotherapy (paclitaxel 135mg/m2 ,iv d1+ carboplatin AUC=5, iv d1), 1 time/3 weeks for 6 weeks, and with intraperitoneal hyperthermic perfusion chemotherapy combined with intraperitoneal cisplatin 40mg/m2，1 time/2 weeks for 6 weeks
  Interventions: Drug: TC:paclitaxel + carboplatin

INTERVENTIONS:
Drug: Bevacizumab
  Arms: Bevacizumab+TC
Drug: TC:paclitaxel + carboplatin

SUMMARY:
To study the efficacy and safety of intraperitoneal injection bevacizumab combined with intraperitoneal hyperthermic perfusion chemotherapy in treatment of malignant ascites of ovarian cancer. To analyze the clinical significance of the concentration change of vascular endothelial growth factor (VEGF) in ascites in treatment of intraperitoneal injection bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patient's awareness and willingness to comply with the study requirements.
* Histologically confirmed and documented ovarian cancer with malignant ascites.
* ECOG(Eastern Cooperative Oncology Group, ECOG) PS 0-2.
* Life expectancy of >3 months.
* No serious inadequate bone marrow function, liver and renal function or significant cardiovascular disease.

Exclusion Criteria:

* Known hypersensitivity to any of the study drugs or excipients.
* Any current anti-cancer therapy.
* No evidence of ascites.
* Key organ dysfunction.
* Significant cardiovascular disease (e.g. congestive heart failure (CHF), uncontrolled cardiac arrhythmia, angina, heart valve disease, myocardial infarction and refractory hypertension need to be long time controlled by medicine).
* Non-healing wound, ulcer or bone fracture.
* Uncontrolled psychiatric history.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 24month

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Hui, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- First Hospital Affiliated to the PLA General Hospital, Beijing,China, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961